CLINICAL TRIAL: NCT06986018
Title: Clinical Study on the Safety, Efficacy, and Pharmacokinetics of a Universal CD19-Targeted CAR-T Cell Injection (RD06-04) in the Treatment of Patients With Refractory Inflammatory Myopathy and ANCA-Associated Vasculitis
Brief Title: Clinical Study on the Targeted CD19 Universal CAR-T Cell Injection (RD06-04) for the Treatment of IIM and AAV
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Director of the Rheumatology and Immunology Department, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD06-04-08
Record Dates: First submitted 2025-04-13; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Inflammatory Myopathies; ANCA-Associated Vasculitis
Keywords: CD19-Targeted Universal CAR-T
MeSH Terms: conditions — Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RD06-04 Cell Injection (Experimental)
  Interventions: Drug: RD06-04 Cell Injection Infusion

INTERVENTIONS:
Drug: RD06-04 Cell Injection Infusion — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

SUMMARY:
This is an open-label, investigator-initiated clinical trial (IIT) designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of RD06-04 in patients with refractory IIM and AAV. The study plans to enroll a total of 12 participants, with 6 cases each for IIM and AAV. Enrollment for both diseases will proceed in parallel. The dose will be 6×10^6 CAR+T cells/kg (±30%), and patients will receive a single infusion of RD06-04.

ELIGIBILITY:
General Inclusion Criteria:

1. The subject voluntarily participates in this trial and has signed the informed consent form.
2. Age ≥18 years and ≤70 years, regardless of gender.
3. Organ Function and Laboratory Tests:

   1. Liver Function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3× upper limit of normal (ULN), total bilirubin (TBIL) ≤2×ULN (except for Gilbert syndrome).
   2. Renal Function: Creatinine ≤1.5×ULN or creatinine clearance ≥40 ml/min.
   3. Blood Routine: Neutrophil count ≥1×10^9/L, hemoglobin ≥60 g/L, platelet count ≥50×10^9/L, lymphocyte count >0.3×10^9/L.
   4. Coagulation Function: International normalized ratio (INR) ≤1.5×ULN, or prothrombin time (PT) ≤1.5×ULN.
   5. Oxygen saturation (SpO2) ≥92% at rest while breathing room air.
   6. Echocardiography shows left ventricular ejection fraction (LVEF) ≥50%.
4. Female subjects of childbearing potential must have a negative serum or urine pregnancy test result during screening.
5. Females of childbearing potential must agree to use highly effective contraception from at least 28 days before the start of lymphodepletion until 12 months after the infusion of RD06-04. Males of reproductive potential must agree to use an effective barrier method of contraception from the start of lymphodepletion until 12 months after the infusion of RD06-04 and must not donate semen or sperm during the entire trial period.

For IIM participants:

1. Diagnosed with IIM (including probable or definite diagnosis, i.e., a probability of ≥55%) according to the 2017 ACR/EULAR classification criteria. Currently, the ENMC considers that the subtypes of IIM mainly include dermatomyositis (DM), antisynthetase syndrome (ASS), and immune-mediated necrotizing myopathy (IMNM).

For AAV participants:

1. Meets the diagnostic criteria for ANCA-associated vasculitis as established by the 2022 ACR/EULAR, including microscopic polyangiitis (MPA), granulomatosis with polyangiitis (GPA), and eosinophilic granulomatosis with polyangiitis (EGPA).

Exclusion Criteria:

1. As determined by the investigator, the primary diagnosis is a rheumatic autoimmune disease other than the disease under study, which the investigator believes may confound the efficacy evaluation of the study disease.
2. Clinically significant central nervous system disease or pathological changes not caused by the non-study disease within 12 months prior to screening.
3. History of allogeneic bone marrow or stem cell transplantation or solid organ transplantation (such as kidney, lung, heart, liver) or plans for such transplantation in the future.
4. For IIM patients: Presence of severe rhabdomyolysis or CK levels ≥120×ULN at screening.
5. History of, or current significant cardiovascular dysfunction.
6. History of malignancy within 5 years prior to signing the ICF.
7. Pregnant or breastfeeding women.
8. History of recurrent infections requiring hospitalization and intravenous antibiotics (e.g., three or more episodes of the same type of infection within the past year).
9. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) with detectable hepatitis B virus (HBV) DNA in peripheral blood; positive for hepatitis C virus (HCV) antibody with detectable HCV RNA in peripheral blood; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis antibody.
10. History of drug or alcohol abuse within 1 year prior to screening.
11. Any condition that, in the investigator's opinion, may affect study participation, pose a safety risk to the patient, or potentially confound the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-14 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (TEAE), Serious Adverse Events (SAE), Adverse Events of Special Interest (AESI) | Up to 2 years

SECONDARY OUTCOMES:
The proportion of patients with kidney involvement achieving complete kidney remission (CRR) | At weeks 12, and months 6, 12, 18, and 24 following CAR-T infusion.
The change in UPCR from baseline in patients with kidney involvement. | At weeks 2, 4, 8, 12, and at months 6, 9, 12, 18, and 24 following CAR-T infusion.
The change in eGFR (estimated glomerular filtration rate) from baseline in patients with kidney involvement. | At weeks 2, 4, 8, 12, and at months 6, 9, 12, 18, and 24 following CAR-T infusion.
The change in BVAS score from baseline in AAV patients | At 6, 12, 18, and 24 months following CAR-T infusion.
  Birmingham Vasculitis Activity Score (BVAS) has a minimum score of 0 and a theoretical maximum score exceeding 100 (depending on the number and severity of affected organ systems).
  A higher score indicates stronger disease activity and a worse prognosis, while a decrease in score (especially to <5) typically suggests effective treatment.
IIM patients were assessed for major clinical remission (Total Improvement Score, TIS) according to the 2016 ACR /EULAR criteria for myocarditis remission. | At 6, 12, 18, and 24 months following CAR-T infusion.
  Total Improvement Score (TIS) has a minimum score of 0 (indicating no improvement) and a maximum score of 100 (indicating maximal improvement).
  A higher score represents more significant disease improvement and better treatment efficacy.
The change in FACIT-Fatigue from baseline. | At 6, 12, 18, and 24 months following CAR-T infusion.
  Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) has a minimum score of 0 and a maximum score of 52.
  A higher score indicates less severe fatigue and better quality of life.
Assessment of the peak amplification level (Cmax), area under the concentration-time curve (AUC0-28), and persistence profile of RD06-04. | Up to 2 years
The change in HAQ-DI from baseline. | At 6, 12, 18, and 24 months following CAR-T infusion.
  Health Assessment Questionnaire-Disability Index (HAQ-DI) has a minimum score of 0 and a maximum score of 3.
  A higher score indicates more severe physical dysfunction and worse quality of life.
Assessment of the incidence and titer levels of anti-RD06-04 specific anti-drug antibodies (ADA). | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No